CLINICAL TRIAL: NCT00761501
Title: Phase I, Open-label, Randomized, 3-way Crossover Study to Assess Relative Bioavailability of Single Oral Dose of Naproxen as PN400 Compared to Naproxen as Proxen S and Naprosyn E in Healthy Volunteers
Brief Title: Phase I Study to Evaluate Bioavailability of Naproxen as PN400 Compared to Naproxen as Proxen S and Naprosyn E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Sostek, MD, Medical Science Director, Development Projects, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D1120C00001
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteer
Keywords: Phase I; Healthy Volunteer
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: PN400
- 2 (Active Comparator)
  Interventions: Drug: Naproxen (Proxen S)
- 3 (Active Comparator)
  Interventions: Drug: Naproxen (Naprosyn E)

INTERVENTIONS:
Drug: PN400 — Oral
  Other Names: VIMOVO™
  Arms: 1
Drug: Naproxen (Proxen S) — Oral
  Other Names: Proxen S
  Arms: 2
Drug: Naproxen (Naprosyn E) — Oral
  Other Names: Naprosyn E
  Arms: 3

SUMMARY:
The purpose of the study is to investigate the uptake in the body of naproxen; one of the two active substances in PN400. We also want to show that the body's uptake of naproxen given as PN400 is comparable to that of currently marketed naproxen tablets.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of greater than or equal to 19 to less than or equal to 30 kg/m2 and weight of greater than or equal to 50 to less than or equal to 100 kg
* Clinically normal physical exams and laboratory measurements

Exclusion Criteria:

* Subject has received another investigational drug within 4 weeks preceding this study or planning to participate in another study at any time during the period of this study
* Any significant medical or psychiatric condition that could affect the interpretation of the PK data, or which otherwise would contraindicate participation in a clinical trial
* Any GI disease, abnormality or gastric surgery that may interfere with gastric emptying, motility and drug absorption
* Subject who has donated a unit of blood or plasma within 3 months prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | pre-dose and multiple times post-dose

SECONDARY OUTCOMES:
Safety | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Aslak Rautio, MD, Principal Investigator — Quintiles Hermelinen; Wolfgang Kuhn, MD, Principal Investigator — Quintiles Phase I Services
Locations (2):
- Sweden (2):
  - Research Site, Luleå
  - Research Site, Uppsala